CLINICAL TRIAL: NCT02824783
Title: Quality of Life and Satisfaction of Patients Discharged Home After Enhanced Recovery Protocol for Colorectal Surgery
Brief Title: Quality of Life After Enhanced Recovery Protocol for Colorectal Surgery
Status: Completed | Type: Observational
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Jean François Brichant, Professor and Chief Department of Anesthesiology, University of Liege
Other Study IDs: GRACE1
Record Dates: First submitted 2016-06-25; First posted 2016-07-07 (Estimated); Last update posted 2018-01-03 (Actual); Status verified 2017-12

CONDITIONS: Surgery
Keywords: colorectal surgery; enhanced recovery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of the study is to investigate the quality of life and satisfaction of patient who underwent colorectal surgery using an enhanced recovery protocol when back home.

In this retrospective study patients will be telephoned and asked to answer a questionnaire.

DETAILED DESCRIPTION:
Since October 1st 2015, our center has been labelled reference center for colorectal surgery using Enhanced Recovery Protocol (ERP) by GRACE (Groupe francophone de Rehabilitation après ChirurgiE; a francophone counterpart of ERAS® society). In case of ERP, the quality of life when the patient is at home is not well known. Some argue that patient might experience discomfort and lack of autonomy, particularly elderly patient if discharged home too quickly.

In this study, the investigators will call our patients introduced in the database of GRACE to assess the quality of life and patient satisfaction concerning our ERP. Eight domains will be investigated: information, stress, feelings when discharged home, pain, fatigue, autonomy, feeding problems, and satisfaction.

When analyzing the results the investigators will pay a particular attention to elderly patients (age > 70 yo) to determine whether these experience more difficulties as compared to younger patients.

ELIGIBILITY:
Inclusion Criteria:

* all patients included in our GRACE database

Exclusion Criteria:

* No exclusion criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: all patients included in our GRACE database since the 1st of October 2015
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2016-01; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Quality of life (0 to ten numeric scale + questionnaire) | first month after leaving the hospital
  0 to ten numeric scale + questionnaire

SECONDARY OUTCOMES:
Satisfaction (0 to ten numeric scale + questionnaire) | first month after leaving the hospital
  0 to ten numeric scale + questionnaire
Pain (0 to ten numeric scale + questionnaire) | first month after leaving the hospital
  0 to ten numeric scale + questionnaire
Fatigue (0 to ten numeric scale + questionnaire) | first month after leaving the hospital
  0 to ten numeric scale + questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Jean Joris, M.D., Principal Investigator — Department of Anesthesiology, CHU Liege, Belgium
Locations (1):
- University Hospital of Liege, Liège, Belgium

IPD SHARING:
Plan to Share IPD: No